CLINICAL TRIAL: NCT07053319
Title: Protocol lV: SGLT2 Inhibitors, Pioglitazone and Ketone Production in Type 2 Diabetes Mellitus
Brief Title: SGLT2i, Pioglitazone, and Ketone Production in T2D
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 20230457HU-504077; R01DK024092 (NIH)
Record Dates: First submitted 2025-06-26; First posted 2025-07-08 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-06

CONDITIONS: Type 2 Diabetes
Keywords: Endogenous glucose production; Ketogenesis; Gluconeogenesis; Lipolysis
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — empagliflozin; Pioglitazone; Sodium-Glucose Transporter 2

STUDY DESIGN:
Intervention Model Description: A randomized controlled 4 arm clinical trial
Who Masked: Participant, Care Provider, Investigator
Masking Description: Subjects will be randomly assigned 1:1:1:1 ratio
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Empagliflozin plus Pioglitazone placebo (Experimental): Empagliflozin 25 mg/day plus pioglitazone placebo
  Interventions: Drug: Empagliflozin 25 MG plus Pioglitazone placebo
- Pioglitazone plus Empagliflozin Placebo (Placebo Comparator): Pioglitazone, 15 mg/day, increased to 30 mg after 2 weeks plus empagliflozin placebo
  Interventions: Drug: Pioglitazone 15 mg increased to 30 mg after 2 weeks plus Empagliflozin Placebo
- Empagliflozin plus Pioglitazone (Experimental): Empagliflozin(25mg/day) plus pioglitazone (15/30 mg/d)
  Interventions: Drug: Empagliflozin 25 mg/d plus Pioglitazone (15/30 mg/d)
- Empagliflozin placebo + pioglitazone placebo (Experimental): empagliflozin placebo plus pioglitazone placebo
  Interventions: Drug: Pioglitazone placebo + Empagliflozin placebo

INTERVENTIONS:
Drug: Empagliflozin 25 MG plus Pioglitazone placebo — A medication used in the management and treatment of type 2 diabetes mellitus. It is in the sodium-glucose co-transporter (SGLT-2) class of medications.
  Other Names: Empagliflozin; Placebo-Inert tablet
  Arms: Empagliflozin plus Pioglitazone placebo
Drug: Pioglitazone 15 mg increased to 30 mg after 2 weeks plus Empagliflozin Placebo — Placebo-Inert tablet
  Other Names: Placebo for empagliflozin; Pioglitazone, a medication used in the management and treatment of type 2 diabetes mellitus. It is in the thiazolidinedione class of medications
  Arms: Pioglitazone plus Empagliflozin Placebo
Drug: Empagliflozin 25 mg/d plus Pioglitazone (15/30 mg/d) — Pioglitazone, a medication used in the management and treatment of type 2 diabetes mellitus. It is in the thiazolidinedione class of medications
  Other Names: Empagliflozin/Pioglitazone; Empagliflozin, a medication used in the management and treatment of type 2 diabetes mellitus. It is in the sodium-glucose co-transporter (SGLT-2) class of medications.
  Arms: Empagliflozin plus Pioglitazone
Drug: Pioglitazone placebo + Empagliflozin placebo — Placebo-Inert tablet
  Other Names: Placebo/Placebo
  Arms: Empagliflozin placebo + pioglitazone placebo

SUMMARY:
To examine whether the empagliflozin-induced stimulation of EGP, lipolysis, and ketone production in T2D individuals can be blocked by pioglitazone (which has direct hepatic and adipose tissue effects).

DETAILED DESCRIPTION:
Participants: 64 T2D subjects with the same inclusion and exclusion criteria as Protocol 1. Subjects with hematuria are excluded.

Study Design: Infusions of 3-3H-glucose and 14C-glycerol are started and continued to study end (2 PM). Baseline blood samples for HbA1c (x2) and for plasma insulin, glucagon, glucose, FFA, BHB, AcAc, glycerol, and plasma 3-3H-glucose and 14C-glycerol specific activities are drawn at -30, -20, -10, -5, and 0 minutes for measurement of lipolysis, ketone production (plasma ketone levels), and EGP. Empagliflozin (25 mg) is ingested at time zero (9AM) and plasma samples for the above are obtained every 10-20 minutes.

Following completion of the above study, subjects will be randomized to one of four groups (16 per group) for 10 weeks: (1) empagliflozin, 25 mg/day, plus pioglitazone placebo; (2) pioglitazone, 15 mg/day, increased to 30 mg after 2 weeks plus empagliflozin placebo; (3) empagliflozin (25 mg/d) plus pioglitazone (15/30 mg/d); (4) empa placebo plus pio placebo. Subjects will return to the CRC every 1-2 weeks for interim medical history, to check medication compliance, and to measure plasma insulin, glucagon, glucose, FFA, glycerol, BHB, and AcAc levels. At week 10, subjects will return to the CRC at 6AM and the baseline study will be repeated. HbA1c will be measured twice during week 10.

ELIGIBILITY:
Patients with T2D

Inclusion Criteria:

* Ages 30-75 years
* Body Mass Index (BMI) 21-45 kg/m2
* Hemoglobin A1C (HbA1c) = 7.0-11%
* Estimated glomerular filtration rate (eGFR) > 60 ml/min/1.73m2
* Blood Pressure (BP) < 145/85 mmHg
* Participants must be in general good health based on medical history, physical exam, screening blood chemistries, complete blood chemistry (CBC), thyroid stimulating hormone/thyroxine (TSH/T4), electrocardiogram (EKG), and urinalysis
* Stable body weight (±1.5 kg) over the last 3 months and must not participate in an excessively heavy exercise program
* Patients treated with diet, sulfonylurea (SU), metformin (MET), or SU/MET
* Statin therapy is permissible if the dose has been stable for at least 3 months

Exclusion Criteria:

* Patients treated with Glucagon-like peptide 1 receptor agonists (GLP-1 RA), Dipeptidyl Peptidase IV inhibitors (DPP-4i), Thiazolidinediones (TZD), or insulin are excluded
* Patients taking medications (other than SU/MET) known to affect glucose metabolism are excluded
* Subjects with evidence of proliferative retinopathy or eGFR < 60 are excluded
* Women of childbearing potential are excluded unless they are taking/using appropriate contractive medications/devices

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Endogenous Glucose Production (EGP) | 0 and 300 minutes
  Measurement of Endogenous Glucose Production (EGP) using stable isotope (6,6, D2- glucose infusion).

CONTACTS AND LOCATIONS:
Overall Officials: Ralph DeFronzo, MD, Principal Investigator — University of Texas Health Science Center San Antonio
Locations (1):
- Texas Diabetes Institute/UH, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data will be shared with NIH and as a publication in a peer reviewed journal once data are published.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: At study end after analysis of data.